CLINICAL TRIAL: NCT04800055
Title: Attractive Targeted Sugar Bait Phase III Trial in Zambia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PATH (Other)
Collaborators: Tulane University (Other); Ministry of Health, Zambia (Other Government); Macha Research Trust, Zambia (Other)
Responsible Party: Principal Investigator, John M. Miller, PhD, Senior Malaria Technical Advisor, PATH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1460046; 1460046-5 (Other: PATH IRBNet)
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Malaria; Malaria,Falciparum; Vector-Borne Transmission of Infection
Keywords: Malaria; Attractive Targeted Sugar Bait; vector control; Africa; Zambia
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Intervention Model Description: An open-label two-arm cluster randomized controlled trial (CRCT) design will be used comparing ATSB + universal coverage with a WHO core vector control intervention vs universal coverage with VC alone (standard of care). Universal VC (mainly LLIN) will be ensured in both arms prior to start of the study and will serve as the standard of care. Arm 1 will receive ATSBs for up to two years. Arm 2 will receive the standard of care of universal vector control coverage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATSB + VC intervention (Experimental): Arm 1 will receive ATSBs for up to two years.
  Interventions: Other: Attractive Targeted Sugar Bait
- VC only (No Intervention): Arm 2 will receive the standard of care of universal vector control coverage.

INTERVENTIONS:
Other: Attractive Targeted Sugar Bait — ATSBs will be installed on all structures of consenting households in intervention areas for six months according to instructions from the manufacturer. Monitoring assistants will be responsible for providing individual level household orientation for the ATSB and seeking informed consent. Prior to ATSB deployment, community sensitization activities will be conducted to prepare communities for the intervention and research activities. Where appropriate, local media may be used to disseminate messages to sensitize the community to the intervention and the research.
  Other Names: ATSB
  Arms: ATSB + VC intervention

SUMMARY:
The trial will evaluate the efficacy of ATSB deployment plus universal coverage of a WHO core vector control (VC) interventions over two transmission seasons on a minimum 30% reduction in cohort clinical disease incidence, confirmed case incidence, and parasite prevalence, as compared with VC alone. Measurement of entomological outcomes, assessment of acceptability and barriers to uptake and consistent use of ATSB, safety and adverse event monitoring and estimation of the cost and cost-effectiveness of ATSB will also occur.

DETAILED DESCRIPTION:
An open-label two-arm cluster randomized controlled trial (CRCT) design will be used comparing ATSB + LLINS vs LLINS alone (standard of care). A cluster trial design is indicated given the intended community-level effect of ATSBs on malaria transmission. Universal LLIN coverage will be ensured in both arms prior to start of the study and will serve as the standard of care. Arm 1 will receive ATSBs for two years. Arm 2 will receive the standard of care of universal LLIN coverage.

Sixty clusters will be used for the trial per site, with 30 clusters allocated to the ATSB intervention plus universal LLIN coverage arm, and 30 clusters allocated to the control with standard of care arm, universal LLIN coverage. Restricted randomization will be used to randomize the 60 clusters to intervention and control arms. The incidence cohort and cross-sectional household surveys will each be powered to detect a 30% reduction in the malaria outcome over two years.

Primary aim:

• Quantify the efficacy of ATSBs for reducing P. falciparum clinical case incidence, parasite prevalence, community infection incidence, and health facility confirmed malaria case incidence.

Secondary aims include:

* Quantify the efficacy of ATSBs for reducing target malaria vector density, altering the population age structure by reducing longevity, and reducing sporozoite and entomological inoculation rates (EIR).
* Assess the durability of the ATSB.
* Assess community acceptance of ATSB.
* Identify barriers to high and effective ATSB coverage.
* Understand the impact of ATSB deployment on LLIN use.
* Document cost and cost-effectiveness of ATSB deployment.

ELIGIBILITY:
Inclusion Criteria:

* Household resident
* ≥12 months and <15 years of age at the time of enrollment
* If age 12 months - 6 years of age, parent or guardian provides consent for child's participant
* If age 7-14 years, parent or guardian provides consent for child's participant and child provides assent for participation

Exclusion Criteria:

* Residence within the buffer zone
* Age <12 months or ≥15 years of age at the time of cohort enrollment
* Household contained a participant in the first cohort (for participation in the second cohort)
* Pregnant at the time of cohort enrollment. Pregnant adolescents are excluded because they are eligible for protection from infection through pregnancy standard of care - intermittent preventative therapy during pregnancy (IPTp), and to avoid undue discomfort with repeated blood sampling.
* Pregnancy at any time during the cohort study. Pregnancy will be identified in adolescents at enrollment and follow-up visits through a single question regarding pregnancy status during each cohort visit. When an adolescent indicates that she is pregnant or is unsure of her pregnancy status, she will no longer be followed for ongoing blood testing for the reasons noted above and will be censored in the analysis.
* Does not provide consent/assent required according to age to participate in the study

Ages: 12 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3480 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical malaria case incidence | Seasonal (6 months)
  Clinical malaria case incidence measured by cohort and defined as fever (history of fever in the past 48 hours or an axillary temperature ≥37.5o C. at follow-up visit) plus a positive RDT in children ≥12 months and <15 years in age.

SECONDARY OUTCOMES:
Time to first infection | Seasonal (6 months)
  Time to first infection measured among the cohort and defined as the time to first PCR infection among participants aged ≥12 months and <15 years of age.
Prevalence, detected by PCR | 6 weeks
  Prevalence of malaria infection measured by the cross-sectional household survey among participants aged ≥6 and older, detected by PCR.
Prevalence, detected by RDT | 6 weeks
  Prevalence of malaria infection measured by the cross-sectional household survey among participants aged ≥6 and older, detected by RDT (patent infection).
Incidence rate of passively reported clinical malaria | Seasonal (6 months)
  Incidence rate of clinical malaria among participants of all ages, defined as the number of malaria confirmed cases (by RDT or microscopy) per 1,000 population per year, using routine data from health facilities linked to study clusters (i.e. by name of village of residence) and cluster population sizes for the denominator.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaoma District, Kaoma, Western Province, Zambia

REFERENCES:
- [Derived] Mancuso B, Orange E, Eisele TP, Ashton RA, Littrell M, Matches M, Miller JM, Chanda J, Assefa S, Wagman J, Silumbe K, Hamainza B, Saili K, Slutsker L, Yukich J. Cost and cost-effectiveness of attractive targeted sugar baits (ATSB) in the context of a phase III cluster randomized control trial in Western Province, Zambia. Malar J. 2025 Dec 19;25(1):54. doi: 10.1186/s12936-025-05716-9. PMID 41420162
- [Derived] Ashton RA, Saili K, Chishya C, Banda Yikona H, Arnzen A, Orange E, Chitoshi C, Chulu J, Tobolo T, Ndalama F, Kyomuhangi I, Ngulube W, Moonga H, Chirwa J, Slutsker L, Wagman J, Chanda J, Miller J, Silumbe K, Hamainza B, Eisele TP, Yukich J, Littrell M. Efficacy of attractive targeted sugar bait stations against malaria in Western Province Zambia: epidemiological findings from a two-arm cluster randomized phase III trial. Malar J. 2024 Nov 15;23(1):343. doi: 10.1186/s12936-024-05175-8. PMID 39548456
- [Derived] Wagman J, Chanda B, Chanda J, Saili K, Orange E, Mambo P, Muyabe R, Kaniki T, Mwenya M, Ng'andu M, Sakala J, Ngulube W, Miller J, Arnzen A, Silumbe K, Mwaanga G, Simubali L, Mungo A, Mburu MM, Simulundu E, Mambwe B, Kasaro R, Mulube C, Mwenda M, Hamainza B, Ashton RA, Eisele TP, Harris AF, Entwistle J, Yukich J, Slutsker L, Burkot TR, Littrell M. Entomological effects of attractive targeted sugar bait station deployment in Western Zambia: vector surveillance findings from a two-arm cluster randomized phase III trial. Malar J. 2024 Jul 18;23(1):214. doi: 10.1186/s12936-024-05045-3. PMID 39026236
- [Derived] Mwaanga G, Ford J, Yukich J, Chanda B, Ashton RA, Chanda J, Munsanje B, Muntanga E, Mulota M, Simuyandi C, Mulala B, Simubali L, Saili K, Simulundu E, Miller J, Hamainza B, Orange E, Wagman J, Mburu MM, Harris AF, Entwistle J, Littrell M. Residual bioefficacy of attractive targeted sugar bait stations targeting malaria vectors during seasonal deployment in Western Province of Zambia. Malar J. 2024 May 29;23(1):169. doi: 10.1186/s12936-024-04990-3. PMID 38811947
- [Derived] Attractive Targeted Sugar Bait Phase III Trial Group. Attractive targeted sugar bait phase III trials in Kenya, Mali, and Zambia. Trials. 2022 Aug 9;23(1):640. doi: 10.1186/s13063-022-06555-8. PMID 35945599